CLINICAL TRIAL: NCT01650298
Title: Pilot Study: Tailored Anticoagulation for Noncontinuous AF
Brief Title: Safety Study on Stopping Anticoagulation Medication in Patients With a History of Atrial Fibrillation
Acronym: TACTIC AF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to slow enrollment.
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 60039204/C
Record Dates: First submitted 2012-07-23; First posted 2012-07-26 (Estimated); Results first posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Pharmaceutical Preparations; Factor Xa Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Remote transmissions were scheduled per each institution's device monitoring protocol. Anticoagulation was initiated/discontinued based on standard of care/guidelines as prescribed by doctor
- Tailored Anticoagulation (TAC) (Experimental): Anticoagulation was initiated or discontinued based on atrial tachycardia / atrial fibrillation (AT/AF) burden as assessed through frequent remote transmissions via Merlin.net.
  Patients sent in biweekly remote transmissions, automatic alert-triggered transmissions for AT/AF burden above a set threshold, and unscheduled patient-activated transmissions as needed
  Interventions: Other: Drug (Direct thrombin or Factor Xa inhibitor)

INTERVENTIONS:
Other: Drug (Direct thrombin or Factor Xa inhibitor) — Patient will stop or restart drug per cardiac device information (AT/AF diagnostics for prespecified AT/AF episode duration per day and total burden).
  Arms: Tailored Anticoagulation (TAC)

SUMMARY:
The purpose of this study is to determine whether it is safe to stop anticoagulation medication in patients with a history of atrial fibrillation (AF) based on information from a pacemaker or implantable cardioverter defibrillator (ICD).

ELIGIBILITY:
Inclusion Criteria:

* Patient has a St Jude Medial device that is compatible with Merlin.net (remote monitoring)
* Patient has history of atrial fibrillation (non-continuous)
* Patient must be taking a a blood thinner medication other than warfarin or aspirin for atrial fibrillation
* Patient is willing to complete a questionnaire

Exclusion Criteria:

* Patient is in atrial fibrillation all of the time
* Patient has a history of stroke or blood clot
* Patient is on warfarin or coumadin
* Patient cannot be taken off of his blood thinner medication due to another medical condition
* Patient is not capable of sending a remote device transmission to doctor once a week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Zimetbaum, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (10):
- United States (10):
  - Jeffrey Goodman, MD, Los Angeles, California
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Sparrow Research Institute, Lansing, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Samaritan Heart and Vascular Institute, Corvallis, Oregon
  - Jefferson Heart Institute, Philadelphia, Pennsylvania
  - Allegheny Singer Research Institute, Pittsburgh, Pennsylvania
  - STAR Clinical Trials, LLC / Cardiology Clinic of San Antonio, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Anticoagulation Taken as Prescribed by Doctor: Anticoagulation presciption will be taken per physician's discretion
- Anticoagulation to be Stopped/Started Per Device Information: Other: The physician will manage the patient's anticoagulation medication by weekly remote monitoring device transmissions
  Drug (Direct thrombin or Factor Xa inhibitor): Patient will stop or restart drug per cardiac device information (AT/AF diagnostics for prespecified AT/AF episode duration per day and total burden).
Period: Overall Study
Arm/Group | Anticoagulation Taken as Prescribed by Doctor | Anticoagulation to be Stopped/Started Per Device Information
Started | 16 | 48
Completed | 11 | 42
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Tailored Anticoagulation: Tailored Anticoagulation (TAC): Anticoagulation to be stopped/started per device information. Patients sent in biweekly remote transmissions, automatic alert-triggered transmissions for AT/AF burden above a set threshold, and unscheduled patient-activated transmissions as needed.
  Drug (Direct thrombin or Factor Xa inhibitor): Patient will stop or restart drug per cardiac device information (AT/AF diagnostics for prespecified AT/AF episode duration per day and total burden).
- Total: Total of all reporting groups
Arm/Group | Control | Tailored Anticoagulation | Total
Number analyzed (Participants) | 16 | 48 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 12 | 15
  >=65 years | 13 | 36 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.0 (11.1) | 71.3 (10.2) | 72.2 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 17 | 23
  Male | 10 | 31 | 41
Region of Enrollment [Number; unit: participants]
  United States | 16 | 48 | 64

OUTCOME MEASURES:

1. Primary Outcome: Total Cumulative Days on Anticoagulation
Description: To assess the reduction in time on anticoagulation, the cumulative total number of days on anticoagulation for each group throughout the follow-up period was determined. This study was designed as a pilot/feasibility study and therefore was not powered to detect thromboembolic events. Per study protocol, all patients completed a 30 day run-in period following enrollment during which anticoagulation could not be stopped regardless of AT/AF burden.
Time Frame: one year
Population: After a 30-day run-in period during which anticoagulation use could not be stopped per study protocol, a total of 14,826 cumulative days of monitoring were completed.
Measure: Number; unit: days on anticoagulation
Groups:
- Control: Anticoagulation medication was per doctor's discretion / standard of care (continuous coagulation)
- Tailored Anticoagulation: Anticoagulation medication was based on patient's AT/AF information from device
Arm/Group | Control | Tailored Anticoagulation
Number analyzed (Participants) | 16 | 48
days on anticoagulation | 5840 | 3763

ADVERSE EVENTS:
Groups:
- Anticoagulation Taken as Prescribed by Doctor: Anticoagulation medication was per doctor's discretion
- Anticoagulation to be Stopped/Started Per Device Information: Anticoagulation medication was based on patient's AT/AF information from device
Arm/Group | Anticoagulation Taken as Prescribed by Doctor | Anticoagulation to be Stopped/Started Per Device Information
All-Cause Mortality (participants affected / at risk) | 0/16 | 2/48
Serious Adverse Events (participants affected / at risk) | 3/16 | 8/48
Other Adverse Events (participants affected / at risk) | 5/16 | 9/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anticoagulation Taken as Prescribed by Doctor (N=16) | Anticoagulation to be Stopped/Started Per Device Information (N=48)
Hemorrahagic event (Gastrointestinal disorders) | 1 (1) | 0 (0) — Patient With Hematemesis And Epigastric Pain. Gi Consult. Egd With Ulcer In Funders Which Was Endoclipped. Continued On Aspirin And Apixaban. Avoid Nsaid.
DECOMPENSATED HF (Cardiac disorders) | 1 (1) | 0 (0)
ATRIAL ARRHYTHMIA (Cardiac disorders) | 1 (2) | 6 (7)
HEMORRHAGIC EVENT (Nervous system disorders) | 0 (0) | 1 (1)
INFECTION (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anticoagulation Taken as Prescribed by Doctor (N=16) | Anticoagulation to be Stopped/Started Per Device Information (N=48)
ATRIAL ARRHYTHMIA (Cardiac disorders) | 1 (1) | 2 (3)
HEMORRHAGIC EVENT (General disorders) | 1 (1) | 0 (0)
HEMORRHAGIC EVENT (Vascular disorders) | 2 (2) | 0 (0)
LV Thrombus (Cardiac disorders) | 1 (1) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HEMORRHAGIC EVENT (Gastrointestinal disorders) | 0 (0) | 2 (2)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1)
DIVERTICULITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
SYNCOPE (General disorders) | 0 (0) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 1 (1)
OVERSENSING (Product Issues) | 0 (0) | 1 (1)
RADIAL HEAD FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No